CLINICAL TRIAL: NCT05268055
Title: Sign Here: How to Conduct Informed Consent With Deaf Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Brown University (Other)
Responsible Party: Principal Investigator, Melissa L. Anderson, Associate Professor of Psychiatry, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: H00021294; 5R21DC019216 (NIH)
Record Dates: First submitted 2022-02-23; First posted 2022-03-07 (Actual); Results first posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Cultural Competency
Keywords: informed consent; simulation; Deaf; cultural competence
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Sign Here" training intervention (Experimental): Participants randomized to the experimental condition will view the new "Sign Here" training film for healthcare providers.
  Interventions: Other: "Sign Here" training intervention
- Intervention as usual (Other): Participants randomized to intervention as usual will review "Communicating with People Who Are Deaf or Hard of Hearing in Hospital Settings" (https://archive.ada.gov/hospcombrprt.pdf)
  Interventions: Other: Intervention as usual

INTERVENTIONS:
Other: "Sign Here" training intervention — Training film to educate healthcare providers to competently and sensitively interact with Deaf patients in healthcare settings.
  Arms: "Sign Here" training intervention
Other: Intervention as usual — "Communicating with People Who Are Deaf or Hard of Hearing in Hospital Settings" (https://archive.ada.gov/hospcombrprt.pdf)
  Arms: Intervention as usual

SUMMARY:
The goal of this research is to create a training film for hearing healthcare providers to teach them how to competently and sensitively interact with Deaf patients. In Year 1, focus groups will be facilitated to elicit feedback that will inform video production of the training film. In Year 2, film production will take place, as well as a randomized clinical trial (RCT) to test the feasibility and preliminary efficacy of the new training intervention.

DETAILED DESCRIPTION:
The U.S. Deaf community - a minority group of more than 500,000 people who use American Sign Language (ASL) - is one of the most understudied and underserved populations within our nation's healthcare system. Reasons for this underrepresentation include lack of language access in healthcare and research settings, as well as communal feelings of mistrust toward the medical community. For example, healthcare providers and clinical researchers follow a medical model to "cure" or "fix" deafness, whereas most Deaf people do not want to be fixed, but rather to be respected as a cultural and linguistic minority group.

To begin to rectify this mistrust and underrepresentation, the informed consent process has been suggested as a key area of intervention. From 2016 - 2018, our team produced a film to train research personnel to effectively interact with Deaf research participants during the informed consent process. The intervention was designed through a two-year collaboration with the local Deaf community - community forums, focus groups, and an intervention development team inclusive of Deaf researchers, filmmakers, and laypeople.

In 2022, our team conducted a second series of focus groups with key stakeholders to refine, expand, and tailor a new version of the Sign Here training film for healthcare providers. Filmmaking is currently underway. In April 2023, we will launch a randomized controlled trial to test the feasibility, acceptability, and preliminary efficacy of the new training intervention. Eighty healthcare providers, medical students, and nursing students will be randomized to receive (1) the Sign Here training film or (2) an "intervention as usual" condition (i.e., standard written guidance on how to communicate with Deaf patients in healthcare settings). Primary outcomes are provider cultural competence, communication skill, and ability to build trust, which will be tested via virtual simulation with a Deaf standardized patient.

Results will potentially validate a product of immediate value - a highly-accessible, easy-to-disseminate training film to promote the inclusion of Deaf people in our nation's healthcare system. Results will also inform the design of a large, multi-institution study to explore the real-world scalability of the Sign Here training film in medical schools across the U.S.

ELIGIBILITY:
Inclusion Criteria:

* age 18+
* self-identification as a healthcare provider, medical student, or nursing student
* current or recent engagement in informed consent for treatment
* access to an informed consent form that can be used for a simulated informed consent session
* We will also screen participants' self-reported level of experience with Deaf people, as we aim to recruit participants with little-to-no prior experience interacting with Deaf people to reflect the most probable real-word encounter that a Deaf person would have when receiving healthcare services.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa L Anderson, Principal Investigator — melissa.anderson@umassmed.edu
Locations (1):
- University of Massachusetts Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 325 healthcare providers, medical students, and nursing students who were screened, 208 met inclusion criteria, consented to participate in the study, and were subsequently randomized to condition. Study participants were either healthcare professionals or students in healthcare professions. The Deaf standardized patient who participated in outcome simulations was a trained member of our research team, not a study participant.
Period: Overall Study
Arm/Group | "Sign Here" Training Intervention | Intervention as Usual
Started | 103 | 105
Reviewed Training Intervention | 51 | 56
Scheduled Study Simulation Session | 35 | 38
Completed Study Simulation Session | 23 | 29
Completed | 23 | 29
Not Completed | 80 | 76
Not completed — Lost to Follow-up | 68 | 68
Not completed — Withdrawal by Subject | 12 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | "Sign Here" Training Intervention | Intervention as Usual | Total
Number analyzed (Participants) | 103 | 105 | 208
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.94 (11.78) | 41.77 (13.48) | 41.36 (12.64)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 85 | 86 | 171
  Gender: Male | 18 | 18 | 36
  Gender: Other | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 14
  Not Hispanic or Latino | 96 | 98 | 194
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 9 | 13 | 22
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 8 | 4 | 12
  White | 84 | 84 | 168
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Healthcare Provider Cultural Competency
Description: A validated scale used to measure provider cultural competence. Total scores range from 9 to 63, with higher scores indicative of higher levels of cultural competency.
Time Frame: post-intervention, up to one month
Population: Enrolled participants who reviewed their assigned training intervention and completed the study simulation session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Sign Here" Training Intervention | Intervention as Usual
Number analyzed (Participants) | 23 | 29
score on a scale
  All participants | 40.5 (14.0) | 42.7 (11.0)
  Participants less than age 33: number analyzed (Participants) | 11 | 15
  Participants less than age 33 | 48.7 (8.3) | 41.3 (9.1)
  Participants aged 33 and greater: number analyzed (Participants) | 12 | 14
  Participants aged 33 and greater | 33.0 (14.2) | 44.3 (13.0)
Statistical Analysis 1: Comparison: "Sign Here" Training Intervention vs Intervention as Usual; Group comparison of all participants; Test type: Superiority; p = 0.525, t-test, 2 sided
Statistical Analysis 2: Comparison: "Sign Here" Training Intervention vs Intervention as Usual; Group comparison of participants less than age 33; Test type: Superiority; p = 0.045, t-test, 2 sided
Statistical Analysis 3: Comparison: "Sign Here" Training Intervention vs Intervention as Usual; Group comparison of participants age 33 and greater; Test type: Superiority; p = 0.046, t-test, 2 sided

2. Primary Outcome: Ask, Understand, Remember Assessment
Description: A validated scale used to measure participants' communication skill. Total scores range from 4 to 16, with higher scores indicating better communication skills.
Time Frame: post-intervention, up to one month
Population: Enrolled participants who reviewed their assigned training intervention and completed the study simulation session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Sign Here" Training Intervention | Intervention as Usual
Number analyzed (Participants) | 23 | 29
score on a scale
  All participants | 12.5 (2.9) | 13.5 (2.2)
  Participants less than age 33: number analyzed (Participants) | 11 | 15
  Participants less than age 33 | 14.4 (1.3) | 13.2 (1.8)
  Participants age 33 and greater: number analyzed (Participants) | 12 | 14
  Participants age 33 and greater | 10.8 (3.0) | 13.7 (2.6)
Statistical Analysis 1: Comparison: "Sign Here" Training Intervention vs Intervention as Usual; Group comparison of all participants; Test type: Superiority; p = 0.200, t-test, 2 sided
Statistical Analysis 2: Comparison: "Sign Here" Training Intervention vs Intervention as Usual; Group comparison of participants less than age 33; Test type: Superiority; p = 0.075, t-test, 2 sided
Statistical Analysis 3: Comparison: "Sign Here" Training Intervention vs Intervention as Usual; Group comparison of participants age 33 and greater; Test type: Superiority; p = 0.015, t-test, 2 sided

3. Primary Outcome: Wake Forest Physician Trust Scale
Description: A validated scale used to measure the ability to build trust with the standardized patient/participant. Total scores range from 10 to 50, with higher scores indicating greater ability to build trust.
Time Frame: post-intervention, up to one month
Population: Enrolled participants who reviewed their assigned training intervention and completed the study simulation session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Sign Here" Training Intervention | Intervention as Usual
Number analyzed (Participants) | 23 | 29
score on a scale
  All participants | 36.4 (9.5) | 39.1 (6.9)
  Participants less than age 33: number analyzed (Participants) | 11 | 15
  Participants less than age 33 | 41.6 (5.2) | 38.4 (5.7)
  Participants age 33 and greater: number analyzed (Participants) | 12 | 14
  Participants age 33 and greater | 31.6 (10.2) | 39.8 (8.2)
Statistical Analysis 1: Comparison: "Sign Here" Training Intervention vs Intervention as Usual; Group comparison of all participants; Test type: Superiority; p = 0.246, t-test, 2 sided
Statistical Analysis 2: Comparison: "Sign Here" Training Intervention vs Intervention as Usual; Group comparison of participants less than age 33; Test type: Superiority; p = 0.151, t-test, 2 sided
Statistical Analysis 3: Comparison: "Sign Here" Training Intervention vs Intervention as Usual; Group comparison of participants age 33 and greater; Test type: Superiority; p = 0.033, t-test, 2 sided

4. Secondary Outcome: Assessment of Intervention Understanding & Retention
Description: A ten-question multiple choice test to assess their understanding and retention of intervention content. Total scores range from 0 to 28, with higher scores indicating greater comprehension and retention.
Time Frame: post-intervention, up to one month
Population: Enrolled participants who reviewed their assigned training intervention and completed the study simulation session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Sign Here" Training Intervention | Intervention as Usual
Number analyzed (Participants) | 23 | 29
score on a scale
  All participants | 22.1 (2.5) | 21.2 (2.7)
  Participants less than age 33: number analyzed (Participants) | 11 | 15
  Participants less than age 33 | 21.9 (1.9) | 21.8 (2.1)
  Participants greater than age 33: number analyzed (Participants) | 12 | 14
  Participants greater than age 33 | 22.3 (3.0) | 20.5 (3.2)
Statistical Analysis 1: Comparison: "Sign Here" Training Intervention vs Intervention as Usual; Group comparison of all participants; Test type: Superiority; p = 0.212, t-test, 2 sided
Statistical Analysis 2: Comparison: "Sign Here" Training Intervention vs Intervention as Usual; Group comparison of participants less than age 33; Test type: Superiority; p = 0.893, t-test, 2 sided
Statistical Analysis 3: Comparison: "Sign Here" Training Intervention vs Intervention as Usual; Group comparison of participants age 33 and greater; Test type: Superiority; p = 0.160, t-test, 2 sided

5. Secondary Outcome: Self-Rating of Simulation
Description: Participants complete a self-assessment using the validated scales described above to rate their conduct of culturally-appropriate informed consent in the simulation and are also asked to provide feedback on the study experience.
  For the Healthcare Provider Cultural Competency scale, total scores range from 9 to 63, with higher scores indicating a better outcome.
  For the Ask, Understand, Remember Assessment, total scores range from 4 to 16, with higher scores indicating a better outcome.
  For the Wake Forest Physician Trust Scale, total scores range from 10 to 50, with higher scores indicating a better outcome.
Time Frame: post-intervention, up to one month
Population: Enrolled participants who reviewed their assigned training intervention and completed the study simulation session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | "Sign Here" Training Intervention | Intervention as Usual
Number analyzed (Participants) | 23 | 29
score on a scale
  Healthcare Provider Cultural Competency (participant self-rating) | 42.6 (5.8) | 41.9 (8.1)
  Ask, Understand, Remember Assessment (participant self-rating) | 12.7 (2.5) | 13.2 (2.1)
  Wake Forest Physician Trust Scale (participant self-rating) | 37.7 (4.3) | 39.9 (4.7)
Statistical Analysis 1: Comparison: "Sign Here" Training Intervention vs Intervention as Usual; Group comparison of self-rating scores on the Healthcare Provider Cultural Competence measure; Test type: Superiority; p = 0.752, t-test, 2 sided
Statistical Analysis 2: Comparison: "Sign Here" Training Intervention vs Intervention as Usual; Group comparison of self-rating scores on the Ask, Understand, Remember Assessment; Test type: Superiority; p = 0.493, t-test, 2 sided
Statistical Analysis 3: Comparison: "Sign Here" Training Intervention vs Intervention as Usual; Group comparison of self-rating scores on the Wake Forest Physician Trust Scale; Test type: Superiority; p = 0.085, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: through study completion, an average of 1 month
Arm/Group | "Sign Here" Training Intervention | Intervention as Usual
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/105
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/15
Other Adverse Events (participants affected / at risk) | 0/103 | 0/105

LIMITATIONS AND CAVEATS:
Small sample size may have affected the power of our statistical analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT05268055/Prot_SAP_000.pdf